CLINICAL TRIAL: NCT06703814
Title: PROtective Ventilation With FLOW-Controlled Ventilation to Improve Postoperative Pulmonary Outcome After ROBOT-Assisted Laparoscopic Surgery - an International Multicenter Pilot Randomized Clinical Trial.
Brief Title: PROtective Ventilation With FLOW-Controlled Ventilation
Acronym: PROFLOW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: University Hospital Bergmannsheil Bochum (Other); Luzerner Kantonsspital (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Dr. Timur Yurttas, MD, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROFLOW-ROBOTic pilot
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pulmonary Complications (PPCs); Feasibility Studies; Pilot Study
Keywords: flow-controlled ventilation; postoperative pulmonary complications; mechanical ventilation; intraoperative ventilation

STUDY DESIGN:
Intervention Model Description: intraoperative Flow-controlled ventilation versus intraoperative pressure-controlled ventilation during general anesthesia
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraoperative flow-controlled ventilation FCV (Experimental): Flow-controlled ventilation (FCV) differs from conventional ventilation modes in several key ways. Unlike pressure-controlled ventilation (PCV) and volume-controlled ventilation (VCV), FCV maintains a constant airflow during both the inspiration and expiration phases. This method generates smooth linear pressure variations by delivering a constant positive flow during inspiration and a constant negative flow during expiration, resulting in linearly changing airway pressures. Additionally, FCV operates without any interruptions in flow throughout the cycle. This consistent rate of pressure and volume change in the lungs, particularly the linear decrease in airway pressure during expiration, has been shown to improve lung recruitment. This approach may thus reduce the risk of pulmonary complications commonly associated with conventional ventilation modes.
  Interventions: Other: Intraoperative flow-controlled ventilation strategy
- Intraoperative pressure-controlled ventilation PCV (Active Comparator): Pressure-controlled ventilation (PCV) is the standard of care in patients undergoing mechanical ventilation during general anesthesia in robot-assisted laparoscopic surgery. The operator sets the inspiratory pressure (rather than tidal volume as in VCV) and respiratory rate (along with FiO2, I:E ratio and PEEP). Typically, the pressure is titrated to achieve a targeted tidal volume.
  Interventions: Other: Intraoperative pressure-controlled ventilation strategy

INTERVENTIONS:
Other: Intraoperative flow-controlled ventilation strategy — In the FCV group, intraoperative ventilation will be provided with the EVONE (IES Ventinova Medical).PEEP and Ppeak are titrated guided by dynamic compliance, as follows: Starting from a default setting of 5 cmH2O of PEEP and 15 cmH2O of Ppeak, PEEP and Ppeak are equally increased by 1 cmH2O steps and the PEEP value with the highest VT and thus highest dynamic compliance is defined as "best" PEEP. Subsequently, Ppeak is stepwise (+1 cmH2O) increased until there is no further over-proportional increase in tidal volume (VT) (i.e. measured VT > expected VT according to measured dynamic compliance), defined as best driving pressure. No recruitment maneuvers are carried out during FCV. With the I:E ratio set to 1:1, flow is adjusted to establish normocapnia (target etCO2 4.5 to 5.8 kPa). FiO2 is adjusted to maintain oxygen saturation (SpO2) > 92%.
  Other Names: FCV
  Arms: Intraoperative flow-controlled ventilation FCV
Other: Intraoperative pressure-controlled ventilation strategy — In the PCV group, intraoperative ventilation will be provided by a standard anesthesia ventilator in use in the respective participating centers. Patients will be ventilated in PCV mode, at the lowest inspired oxygen fraction (FiO2), to maintain oxygen saturation (SpO2) > 92%. It is left to the discretion of the attending anesthesiologist to use a higher fraction of FiO2. Inspiratory to expiratory ratio is set at 1:1 to 1:2, respiratory rate will be adjusted to target normocapnia (target etCO2 4.5 to 5.8 kPa. VT will be set at 7 to 9 ml/kg predicted body weight (PBW). The PBW is calculated according to a predefined formula: 50 + 0.91 x (centimeters of height - 152.4) for males and 45.5 + 0.91 x (centimeters of height - 152.4) for females. Ventilation starts with 5 cm H2O PEEP, and can be increased to 10 cm H2O PEEP.
  Other Names: PCV
  Arms: Intraoperative pressure-controlled ventilation PCV

SUMMARY:
The investigators want to investigate in patients undergoing robot-assisted laparoscopic surgery (a minimally invasive procedure) how applicable flow-controlled ventilation is, and whether it might also be safer than the current ventilation techniques, as well as its impact on potentially reducing the risk of lung-specific complications.

Flow-controlled ventilation has already been tested in several studies on animals and humans and has proven to be a safe form of ventilation for patients undergoing surgery under general anesthesia.

When patients undergo major surgery, general anesthesia is required and, as a result, mechanical ventilation of the lungs. Especially in long and complex surgeries, ventilation can become more difficult or lead to complications postoperatively. These patients may then experience shortness of breath, coughing, or require medication to improve lung function. In some cases, reintubation or additional mechanical ventilation may be necessary for support.

Previous human studies have shown that flow-controlled ventilation is less stressful and, therefore, potentially safer for the lungs compared to traditional ventilation techniques, and that less supplemental oxygen is required. This effect and the safety of flow-controlled ventilation have been demonstrated in several studies.

Therefore, in this study, the investigators aim to explore whether flow-controlled ventilation is potentially safer and easier to apply than traditional ventilation techniques and whether it can reduce the risk of lung-specific complications following robot-assisted surgeries, thereby improving the recovery process postoperatively.

DETAILED DESCRIPTION:
The optimization of intraoperative ventilation is important in patients under general anesthesia, when physiologic breathing is replaced by non- physiologic artificial ventilation. Especially in patients undergoing robot- assisted laparoscopic surgery, intraoperative ventilation can be challenging, because of changes in compliance of the respiratory system and associated problems in gas exchange, due to the pneumoperitoneum and often extreme body positioning. Intraoperative lung-protection strategies have steadily improved in recent years to reduce complications from mechanical ventilation, but postoperative pulmonary complications remain a risk factor for increased morbidity and mortality. This pilot trial will be conducted to evaluate the safety and feasibility of intraoperative FCV during robot-assisted laparoscopic abdominal, urologic, or gynecologic surgery, and will inform the design of a future trial that will test the efficacy of intraoperative FCV compared to PCV in these patients. In an international multicenter randomized clinical pilot trial, intraoperative flow-controlled ventilation (FCV) will be compared with pressure-controlled ventilation (PCV) in patients scheduled for robot-assisted laparoscopic abdominal, urologic, or gynecologic surgery. This pilot trial is designed to test the safety and feasibility of FCV, and to inform the design of a future trial testing the efficacy of FCV with regard to postoperative outcomes, including postoperative pulmonary complications. The ventilation modes are conducted with CE-marked medical devices (anesthesia ventilators or medical ventilators), however these medical devices themselves are not under investigation. All CE-marked standard medical devices from varied manufacturers in use at the participating study centers will be used in full accordance with the instructions for use.

Given that ventilation strategies inherently carry certain risks, yet remain essential in the context of general anesthesia and surgery, it is ethically justified to first conduct a pilot trial. The potential benefits of FCV are significant and warrant investigation. Therefore, the investigators find it appropriate to compare FCV with existing strategies such as PCV, as the investigators anticipate meaningful improvements in patient outcomes with minimal additional risk.

The investigators hypothesize, that FCV is a safe and feasible ventilation strategy in patients undergoing robot-assisted laparoscopic surgery.

The primary objective of this study is to evaluate the safety of intraoperative FCV in patients undergoing robot-assisted laparoscopic surgery, with a focus on: gas exchange, including both oxygenation and decarboxylation; minute ventilation, during all phases of intraoperative ventilation; key ventilator settings and ventilation parameters; respiratory complications, including pneumothorax and hemodynamic complications, including hypotension and arrhythmias.

The secondary objectives are to assess the feasibility of intraoperative FCV and the study protocol in patients undergoing robot-assisted laparoscopic surgery, including an evaluation of the use of FCV. The need for rescue ventilation strategies, i.e., whether FCV (as well as PCV) can be used during all phases of intraoperative ventilation; and compliance with the study protocol, omissions in the eCRF, and the feasibility of follow-up, i.e., how well each PPC can be captured.

The explorative secondary objective concerns the primary endpoint of a future randomized clinical trial testing the efficacy of FCV, i.e., its effects on postoperative pulmonary complications. Herein the investigators will determine the exact incidence, and define the effect size of the intervention.

The primary endpoint of this pilot trial is a set of safety parameters for FCV, including: gas exchange: (hourly) PaO2, PaCO2, SpO2 and end-tidal CO2; minute ventilation: (hourly) total minute volume; ventilator settings and ventilation parameters: (hourly) tidal volume, respiratory rate, PEEP and PIP, FiO2, driving pressure and mechanical power of ventilation, and respiratory system compliance and elastance; intraoperative respiratory complications: (any time point) pneumothorax. intraoperative hemodynamic complications: (any time point) occurrence of hypotension, defined as a mean arterial pressure (MAP) below 65 mm Hg, lasting longer than 1 minute (not related to the surgical course or anesthetic interventions, according to the attending anesthesiologist); and (hourly) vasopressor support and dose; and (any time point) occurrence of arrhythmias, and intervention for arrhythmias.

Secondary endpoints focus on evaluating the feasibility of intraoperative FCV and the study protocol, including: ventilation protocol adherence; and study protocol adherence; and completeness of the eCRF and follow-up of PPCs.

The explorative secondary endpoint will compare FCV with PCV ventilation with respect to predefined and previously used postoperative (pulmonary) complications in the first seven postoperative days, including: mild respiratory failure, defined as the occurrence of one or multiple of the following conditions after more than two days postoperatively: the occurrence of oxygen saturation (SpO2) < 90% or partial pressure of oxygen in the arterial blood (PaO2) < 7.9 kPa (or < 50 mm Hg) on room air, but responding to supplemental oxygen; or a sudden increase in supplemental oxygen requirement to maintain adequate saturation (SpO2 > 90%) in patients receiving routine postoperative oxygen therapy; or any level of supplemental oxygen; severe respiratory failure, defined as need for noninvasive or invasive mechanical ventilation, or a PaO2 < 60 mm Hg (or < 7.9 kPa) or SpO2 <90% despite supplemental oxygen in spontaneously breathing patients; dyspnea, defined as the patient's perception of an uncomfortable abnormal awareness of breathing or respiratory limitation (shortness of breath, inability to take a deep breath, or chest tightness); productive cough, defined as cough that produces sputum or mucus; bronchospasm, defined as newly detected expiratory wheezing treated with bronchodilators; suspected pulmonary infection, defined as receiving antibiotics and meeting at least one of the following criteria: new or changed sputum, new or changed lung opacities on chest radiograph when clinically indicated, tympanic temperature > 38.3°C, white blood cell count > 12,000/μL; pulmonary infiltrate, defined as any unilateral or bilateral infiltrates on chest radiography; aspiration pneumonitis, defined as respiratory failure after the inhalation of regurgitated gastric contents; atelectasis, defined as lung opacification with shift of the mediastinum, hilum, or hemidiaphragm towards the affected area, and compensatory overinflation in the adjacent non-atelectatic lung on chest radiography; ARDS (according to the new global definition of ARDS); pleural effusion, defined as blunting of the costophrenic angle, loss of the sharp silhouette of the ipsilateral hemidiaphragm in upright position, evidence of displacement of adjacent anatomical structures or (in supine position) a hazy opacity in one hemithorax with preserved vascular shadows on chest radiography; pneumothorax, defined as air in the pleural space with no vascular bed surrounding the visceral pleura on chest radiography; cardiopulmonary edema, defined as clinical signs of congestion, including dyspnea, edema, rales and jugular venous distention, with the chest radiograph demonstrating increase in vascular markings and diffuse alveolar interstitial infiltrates; and death in hospital (defined as death from any cause during hospitalization)

The patient population will be selected by the following criteria:

Inclusion criteria: aged ≥ 18 years; and scheduled for elective robot-assisted laparoscopic abdominal, urologic or gynecologic surgery in supine or Trendelenburg position; AND with an increased risk of PPC, according to the ARISCAT risk score (≥ 26 points); OR the combination of age > 40 years, scheduled surgery lasting > 2 hours and planned to receive an intra-arterial catheter for blood pressure monitoring during the surgery; and able to give written informed consent.

Exclusion criteria: body weight < 40 kg; ASA Physical Status Classification System score IV - VI; previous enrolment in the current study; being the study investigator of this study, his/her family members, employees and other dependent persons; known pregnancy or a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating; or no written informed consent.

The sample size calculation is based on the following assumption:

To estimate the appropriate sample size for this pilot trial, the investigators considered both safety and feasibility across multiple centers. Assuming a target of 10 to 15 participants per randomization group in each of the four centers, the total sample size would range from 80 to 120 participants (4 centers × 10-15 participants × 2 randomization groups). For practical purposes and to ensure a robust assessment of the trial's objectives, the investigators have selected a total sample size of 100 participants. This number balances logistical feasibility with the need for adequate data to assess safety outcomes.

The statistical analysis will be performed accordingly. Balance between study groups will be ensured by randomization and an appropriate sample size. Baseline characteristics will be assessed by appropriate tests to demonstrate balance between groups. The investigators will primarily perform an intention to treat analysis, and will add a per protocol analysis as sensitivity analysis. Tests for normal distribution of the data will include QQ-plot assessments. Potential differences between the two groups in the distribution of dichotomous data are analyzed by chi-square statistics.

Continuous data are analyzed by parametric (t-test, ANOVA) or non-parametric (Mann-Whitney U) test for unpaired comparison as appropriate. A sub-analysis related to sex, age, type of surgery will be performed for all study endpoints.

Datasets to be analyzed, analysis populations All participants will be analyzed in terms of the respective endpoint parameters. The data of patients who leave the study prematurely are analyzed independently of the completion of the study (intention to treat). A subgroup analysis with respect to sex, age, type of surgery will be performed for all study endpoints.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective robot-assisted laparoscopic surgery in supine or Trendelenburg position (either abdominal, urologic or gynecologic surgery);
* AND increased risk of PPCs according to the ARISCAT risk score (≥ 26 points);
* OR the combination of age > 40 years, scheduled surgery lasting > 2 hours and planned to receive an intra-arterial catheter for blood pressure monitoring during the surgery;
* aged ≥ 18 years; and
* able to give written informed consent to participate in the study and agree to comply with the study protocol prior to initiation of any study-mandated procedure and study intervention.

Exclusion Criteria:

* ideal body weight < 40 kg;
* ASA Physical Status Classification System score IV - VI;
* previous enrolment into the current study;
* being the study investigator, his/her family members, employees and other dependent persons;
* if female and of childbearing potential, known pregnancy or a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating; or
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of intraoperative FCV | After induction of general anesthesia and beginning of intraoperative mechanical ventilation to the end of surgery and the end of mechanical ventilation (up to a duration of 12 hours of mechanical ventilation).
  The primary objective of this pilot trial is to evaluate the safety of intraoperative FCV in patients undergoing robot-assisted laparoscopic surgery.
  Herein the investigators focus on, gas exchange, including both oxygenation and decarboxylation; minute ventilation, during all phases of intraoperative ventilation; key ventilator settings and ventilation parameters; respiratory complications, including pneumothorax and hemodynamic complications, including hypotension and arrhythmias.

SECONDARY OUTCOMES:
feasibility of intraoperative FCV, study protocol and database completeness | After induction of general anesthesia and beginning of intraoperative mechanical ventilation to the seventh postoperative day or until end of hospitalization, whatever comes first (i.e., up to 7 days after surgery)
  Secondary objectives of this pilot trial are to assess the feasibility of intraoperative FCV in patients undergoing robot-assisted laparoscopic surgery, the feasibility of the study protocol and its electronic case report form (eCRF).
  Herein the investigators focus on: the need for rescue ventilation strategies, i.e., whether FCV (as well as PCV) can be used during all phases of intraoperative ventilation; and compliance with the study protocol, omissions in the eCRF, and the feasibility of follow-up, i.e., how well each postoperative pulmonary complication can be captured.

OTHER OUTCOMES:
Explorative objective incidence of PPC | After induction of general anesthesia and beginning of intraoperative mechanical ventilation to the seventh postoperative day or until end of hospitalization, whatever comes first (i.e., up to 7 days after surgery)
  Another secondary objective concerns the primary endpoint of a future randomized clinical trial testing the efficacy of FCV, i.e., its effects on postoperative pulmonary complications. Herein the investigators will focus on: the incidence of PPCs in the FCV group and the PCV group, to inform the sample size calculation of the future trial.

CONTACTS AND LOCATIONS:
Overall Officials: Timur Yurttas, MD, Principal Investigator — Department of Anesthesiology, Rescue- and Painmedicine, Cantonal Hospital St. Gallen, Switzerland
Locations (4):
- Department of Anesthesiology, Intensive Care and Pain Medicine, BG University Hospital Bergmannsheil, Ruhr-University Bochum, Germany, Bochum, Germany, Germany
- Department of Anesthesiology, Amsterdam UMC, Amsterdam, Netherlands
- Switzerland (2):
  - Department of Anesthesiology, Cantonal Hospital Luzern, Lucerne, Canton of Lucerne
  - Department of Anaesthesiology, Rescue- and Pain Medicine Cantonal Hospital St. Gallen, Sankt Gallen, Canton of St. Gallen

IPD SHARING:
Plan to Share IPD: No